CLINICAL TRIAL: NCT00689026
Title: Efficacy of Lubiprostone Used With Polyethylene Glycol to Enhance Colonoscopy Preparation Quality in Diabetic Patients: A Randomized Single-Blind Controlled Trial
Brief Title: Efficacy of Lubiprostone in Combination With Standard PEG Preparation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Augusta University (Other)
Collaborators: Takeda Pharmaceuticals North America, Inc. (Industry)
Responsible Party: Principal Investigator, Sherman Chamberlain, Associate Professor, DOM - Gastroenterology, Augusta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: MCG 08-02-186
Record Dates: First submitted 2008-05-29; First posted 2008-06-03 (Estimated); Results first posted 2014-10-20 (Estimated); Last update posted 2014-10-20 (Estimated); Status verified 2014-10

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
Keywords: Colonoscopy; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Cleansing; Preparation; PEG; Quality
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — Lubiprostone; Polyethylene Glycols; Electrolytes; polyethylene glycol 3350

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental (Experimental): The lubiprostone group will receive an additional two 24 mcg lubiprostone capsules, which will be taken orally the morning and evening of the day of the 4L PEG prep (before and after the 4L PEG prep).
  Interventions: Drug: Lubiprostone; Other: Polyethylene glycol with electrolytes
- Control (Active Comparator): All patients in the study will receive a standard oral dosing of 4L Polyethylene glycol with electrolytes colonoscopy preparation the day prior to their scheduled colonoscopy.
  Interventions: Other: Polyethylene glycol with electrolytes

INTERVENTIONS:
Drug: Lubiprostone — Two 24 mcg lubiprostone capsules, which will be taken orally the morning and evening of the day of the 4L PEG prep (before and after the 4L PEG prep).
  Other Names: Amitiza
  Arms: Experimental
Other: Polyethylene glycol with electrolytes — Standard oral dosing of 4L Polyethylene glycol colonoscopy preparation the day prior to their scheduled colonoscopy.
  Other Names: PEG; Nulytely

SUMMARY:
A large population-based study has shown diabetes to be an independent risk factor for colon cancer compared to the general population. Thus, the completion of an adequately prepped colonoscopy is requisite in providing diabetics with adequate colon cancer screening.

Recent data has shown that diabetic patients have poorer response to bowel cleansing compared to non-diabetics (with a standard PEG prep, only 62% of diabetic patients had their colonoscopy preps rated as good or better vs. 97% of normal patients, p<0.001). This may be due to the fact that a majority of diabetic patients report constipation as a common gastrointestinal complaint.

We postulate that lubiprostone (Amitiza), in combination with PEG, will have additional efficacy over standard PEG preparation, and provide optimal safe and effective colonic cleansing for diabetics.

DETAILED DESCRIPTION:
STUDY DESIGN

This is an investigator-initiated, single site (MCG only), single-blinded prospective study comparing the efficacy of Lubiprostone and 4L PEG (Nulytely) to 4 Liters (4L) PEG alone on preparation quality in patients with known diabetes undergoing colonoscopy. Diabetic outpatients who require a colonoscopy will be randomized to one of the two groups of 60 (total of 120 patients):

Control Group: All patients in the study will receive a standard oral 4L PEG colonoscopy preparation the day prior to their scheduled colonoscopy.

Lubiprostone Group: The lubiprostone group will receive an additional two 24 mcg lubiprostone capsules, which will be taken orally the morning and evening of the day of the 4L PEG prep (before and after the oral 4L PEG preparation).

Randomization Scheme: Subjects will be assigned to the Control Group or Lubiprostone Group, on an odd/even basis. After research informed consent has been obtained, subjects are given a study Identification (ID) numbered 1 through 120. Subjects with an odd number will be assigned to Control Group, and subjects with an even number will be assigned to the Lubiprostone Group. Subjects then will be given a randomization package consisting of the preparation orders, supplies, instructions and the date of their procedure by the investigator obtaining informed consent. The colonoscopist will be blinded to which preparation was given.

Only diabetic patients who require an outpatient colonoscopy by a gastroenterologist at the outpatient MCG Clinic will be eligible for the study. Patients will be presented with a separate consent form for the colonoscopy procedure itself.

Standard of Care Procedures

* Colonoscopy Procedure Consent
* Colonoscopy

Study Procedures

* Research Informed Consent
* Disbursement of randomized preparation order and supplies, instructions, and date of procedure to subjects
* Adverse Events

After the procedure, the physician who performed the colonoscopy will complete a form that rates the quality of the subject's colonoscopy preparation on a 1-5 rating scale.

The subject's study participation duration is two days (day of preparation and day of procedure). No follow-up visits will occur.

ELIGIBILITY:
Inclusion Criteria:

* Patients with known diabetes (type I or II) undergoing elective colonoscopy at the Medical College of Georgia.
* Patients aged 50 years and older.
* Women must be post-menopausal or surgically sterile.
* Patients able to give a valid, informed consent.

Exclusion Criteria:

* Patients with impaired glucose tolerance.
* Patients with suspected acute or chronic pseudo-obstruction.
* Patients with active gastrointestinal bleeding.
* Patients with known inflammatory bowel disease.
* Patients with chronic diarrhea.
* Patients with prior colonic resection.
* Patients with active diverticulitis.
* Patients with a known colonic mass.
* Patients with clinical evidence of decompensated liver disease.
* Patients with clinical evidence of decompensated renal disease or patients on dialysis.
* Patients currently or previously taking lubiprostone.
* Patients with an allergy to lubiprostone.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-05; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sherman M Chamberlain, MD, Principal Investigator — Augusta University
Locations (1):
- Medical College of Georgia, Augusta, Georgia, United States

REFERENCES:
- [Result] Grigg E, Schubert MC, Hall J, Rahhal F, Raina D, Sridhar S, Chamberlain SM. Lubiprostone used with polyethylene glycol in diabetic patients enhances colonoscopy preparation quality. World J Gastrointest Endosc. 2010 Jul 16;2(7):263-7. doi: 10.4253/wjge.v2.i7.263. PMID 21160617

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participation was offered to all adult-onset diabetic outpatients 50 and over who were referred to the Gastroenterology clinic at the Medical College of Georgia in Augusta, Georgia for a screening colonoscopy from July, 2008 to March, 2010.
Groups:
- Experimental: Experimental group received one dose of polyethylene glycol electrolyte (PEG) and one does of lubiprostone two hours prior to and two hours after PED completion on the evening prior to the colonoscopy.
- Control: Control group received the standard treatment of polyethylene glycol electrolytes the evening prior to the colonoscopy.
Period: Overall Study
Arm/Group | Experimental | Control
Started | 30 | 30
Completed | 17 | 24
Not Completed | 13 | 6
Not completed — Withdrawal by Subject | 13 | 6

BASELINE CHARACTERISTICS:
Groups:
- Experimental: PEG plus lubiprostone colon cleansing
- Control: PEG colon cleansing
- Total: Total of all reporting groups
Arm/Group | Experimental | Control | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 30 | 60
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (7) | 62 (8) | 58.5 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 17 | 35
  Male | 12 | 13 | 25
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Patients That Received a Quality of Colonoscopy Preparation Rating of <=2 on a 5 Point Likert Scale.
Description: The quality of colonoscopy preparations as rated by blinded colonoscopists on a 5-point Likert Scale where 1=excellent, 2=good, 3=fair, 4=poor, 5=inadequate. It was expected that at least 100 patients would complete the trial.
Time Frame: The outcome was measured at the completion of the colonscopy procedure. Average time to completion two hours
Population: 13 patients were excluded from the Experimental Arm (12 cancelled their appointment and 1 did not complete the prep) and 6 were excluded from the Control Arm (5 cancelled their procedure and 1 withdrew from the trial) therefore results were analyzed and compared using the chi-square statistics-Validated Aronchik colonoscopy cleansing grading scale.
Measure: Number; unit: percentage of patients
Groups:
- Experimental: Lubiprostone: Two 24 mcg lubiprostone capsules, which will be taken orally the morning and evening of the day of the 4 Liters PEG prep (before and after the 4 Liters PEG prep).
- Control: All patients in the control will receive a standard oral 4 Liters PEG colonoscopy preparation the evening prior to their scheduled colonoscopy.
Arm/Group | Experimental | Control
Number analyzed (Participants) | 17 | 24
percentage of patients | 47 | 25

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Treatment: Patients who were given a two doses of lubiprostone with the PEG colon cleansing solution on the day prior the recorded colonoscopy for cleansing grading
- Control: Patients received a standard oral 4 Liters PEG colonoscopy preparation the evening prior to their scheduled colonoscopy
Arm/Group | Treatment | Control
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/24
Other Adverse Events (participants affected / at risk) | 1/17 | 0/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=17) | Control (N=24)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0) — Subject given lubiprostone was found to have an isolated event of atrial fibrillation on presentation for colonoscopy. This was determined to be an unrelated, incidental, adverse event and reported to the Institutional Review Board of record.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No